CLINICAL TRIAL: NCT06625281
Title: Effects of Epleys Maneuver Versus Semont-Plus Maneuver Combined with Brandt-Daroff Exercises on Dizziness and Quality of Life in Benign Paroxysmal Positional Vertigo;
Brief Title: Effects of Epleys Maneuver Versus Semont-Plus Maneuver Combined with Brandt-Daroff Exercises on Dizziness and Quality of Life in Benign Paroxysmal Positional Vertigo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/30
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Dizziness; Benign Paroxysmal Positional Vertigo (BPPV)
Keywords: PhysicalTherapy; Vestibular Rehabilitation Therapy; Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Dizziness; Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be kept unaware of which group they will be allocated and type of the intervention they will receive, whereas the investigator will be aware regarding the allocation and type of the intervention given to the participants. Single blinding is used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group A (Active Comparator): It includes participants receiving Epley's Maneuver combined with Brandt-daroff exercises for 6 weeks of treatment.
  Interventions: Procedure: Epleys Maneuver; Procedure: Brandt-Daroff exercises
- Interventional Group B (Experimental): This group involves participants receiving Semont-Plus Maneuver along with Brandt-daroff exercises for a period of 6 weeks.
  Interventions: Procedure: Semont-plus maneuver; Procedure: Brandt-Daroff exercises

INTERVENTIONS:
Procedure: Epleys Maneuver — * The patient begins in an upright sitting posture, with the legs fully extended and the head rotated 45 degrees towards the affected side.
  * The patient is then quickly and passively forced down backwards by the therapist performing the treatment into a supine position with the head held approximately in a 30-degree neck extension
  * The therapist observes the patient's eyes for "primary stage" nystagmus. The patient remains in this position for 1-2 minutes.
  * The patient's head is then turned 90 degrees to the opposite direction so that the unaffected ear faces the ground, for 1-2 minutes.
  * Keeping the head and neck in a fixed position relative to the body, the individual rolls onto their shoulder, rotating the head another 90 degrees in the direction they are facing. The patient is now looking downwards at a 45-degree angle.
  * The eyes should be immediately observed by the therapist for "secondary stage" nystagmus. The patient remains in this position for 1-2 minutes.
  Arms: Interventional Group A
Procedure: Semont-plus maneuver — * The Semont-plus maneuver includes the upright position with turning of the head by 45° toward the non-affected side.
  * Then movement of the body by 150° toward the affected side, which moves the otoconia further in the direction in which they should move and since the clot is beyond the vertex, the movement of body by 240° moves the clot into the direction of the vestibulum.
  Arms: Interventional Group B
Procedure: Brandt-Daroff exercises — * Patient sits on the edge of bed. and lies down onto the side that causes dizziness to increase. Look towards the ceiling. Stay in this position for 2 minutes.
  * Sits upright and then wait for 30 seconds.
  * Moves rapidly to the opposite side for 2 minutes.

SUMMARY:
Vestibular hypofunction can result in symptoms consisting of dizziness, imbalance, and/or oscillopsia, gaze and gait instability, and impaired navigation and spatial orientation; thus, may negatively impact an individual's quality of life, and ability to perform activities of daily living.

Benign paroxysmal positional vertigo (BPPV) is the most common peripheral vestibular disorder which occurs with changing of the positions lying down, rolling over, climbing stairs, or looking up and down. The typical symptoms include dizziness, loss of balance, nystagmus, and nausea, limiting the daily activities of life and functional capacity.

Much research has been done to rule out the prime treatment for posterior canal-BPPV using vestibular rehabilitation therapy (VRT), Canalith repositioning maneuvers (CRM), and habituation exercises, but scarce literature renders the combination of maneuvers and exercises.

The current study will be used to determine and compare the effects of Epley's maneuver Versus the Semont-Plus maneuver combined with Brandt-Daroff exercises on Dizziness and Quality of life in participants with pc-Benign paroxysmal positional vertigo. The participants having clinically diagnosed Posterior canal Benign paroxysmal positional vertigo (BPPV) will be selected in this study.

The outcome measure will be the Dizziness Handicap Inventory (DHI) to assess the Dizziness in participants and Vestibular activities and the participation measure (VAP) will assess the Quality of life. For such a randomized control trial a sample of 40 participants will be taken with 20 participants in each group will be included in the study. One group will undergo Epley's Maneuver and Brandt-daroff exercises and the second group will receive Semont-plus maneuver and Brandt-daroff exercises. Scores will be taken again after intervention. The study will be conducted over 1 year at Fauji Foundation Hospital and Foundation University Islamabad. Participants of interest would be approached and explained about the research. Informed written consent will be taken first. Recruited participants will be allocated to either of the groups through a convenient sampling method.

All outcome measurements would be performed first at baseline and then after the 6 weeks intervention period..

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the Effects of Semont-Plus Maneuver combined with Brandt-Daroff exercises on Dizziness and Quality of life in patients with pc-Benign paroxysmal positional vertigo (BPPV) 2-To determine the Effects of Epley's Maneuver combined with Brandt-Daroff exercises on dizziness and Quality of life in patients with pc-Benign paroxysmal positional vertigo (BPPV) 3-To compare the effects of Epley's maneuver combined with Brandt-daroff exercises with the effects of Semont plus maneuver combined with Brandt-daroff exercises on Dizziness and Quality of life in patients with pc-Benign paroxysmal positional vertigo (BPPV)

HYPOTHESIS:

Alternate Hypothesis:

There will be a significant effect in the study group in terms of Dizziness and Quality of life between Epley's maneuver combined with brandt-daroff exercises Versus Semont-plus maneuver combined with Brandt-Daroff exercises in patients with pc-BPPV (p<0.05).

Null Hypothesis:

1. There will be no significant effect in the study groups in terms of Dizziness and Quality of life between Epley's maneuver combined with brandt-daroff exercises Versus Semont-plus maneuver combined with Brandt-Daroff exercises in patients with pc-BPPV (p>0.05).

Research Design: Experimental study. Randomized Control Trial

Clinical setting: ENT Department, Fauji Foundation Hospital and Treatment room FUCP.

Study duration: 6 months

Selection Criteria:

Inclusion Criteria

1. Both genders
2. Positive Dix Hallpike test.
3. Patients diagnosed with Posterior canal Benign Paroxysmal Positional Vertigo.
4. Patients with recurrent episodes of dizziness.
5. Age group 20-65.
6. Positive Dix Hallpike Test

Exclusion Criteria

1. Dix Hallpike test negative.
2. DHI Scale: 54+ Severe
3. Trauma
4. Ankylosing spondylitis
5. Cervical pathology-related dizziness
6. Spinal cord injury
7. Carotid stenosis
8. Other Vestibular pathologies (Meniere's disease, Vestibular hypofunction, Labyrinthitis

Sampling technique: Convenience Sampling

Outcome Measures:

Data will be collected on Demographics and general information. Dizziness will be assessed through the Dizziness Handicap Inventory (DHI) and Quality of life will be recorded with a Vestibular assessment and participation measure (VAP).

Experimental Group (A) = This group will receive Semont-Plus Maneuver combined with Brandt-daroff exercises interferential therapy and strengthening exercises and their outcomes will be measured at baseline and at the end of 6 weeks of treatment.

Control group (B) =This group will undergo Epley's maneuver combined with Brandt-daroff exercises their outcomes will be observed at the baseline and then after treatment of 06 weeks.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data will be analyzed based on the study design chosen which is a random control experimental study within the community.

A printed questionnaire will be provided to the patients after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

1. Semont-Plus maneuver is a modified form of the Semont maneuver which has been more effective for posterior canal-related vertigo. It is important to find more evidence regarding the Semont-plus maneuver and Brandt-daroff habituation exercises. The combination of this maneuver with Brandt-Daroff exercises will have a remarkable effect on dizziness and thus improve the quality of life of the patients.
2. This study will provide valuable data regarding the comparison of Epley's Maneuver and Semont Maneuver along with their combination with Brandt-daroff exercises.
3. This study will provide awareness and valuable literature regarding the comparison and combination of maneuvers and exercises. Scarce literature is present regarding the combination of vestibular maneuvers and exercises.
4. An awareness for the health care community to use a new technique of combination. The maneuvers and exercises are quick to perform and can be a part of clinical and emergency conditions.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Positive Dix Hallpike test.
* Patients diagnosed with Posterior canal Benign Paroxysmal Positional Vertigo.
* Patients with recurrent episodes of dizziness.
* Age group 20-65.
* Positive Dix Hallpike Test

Exclusion Criteria:

* Dix Hallpike test negative.
* DHI Scale: 54+ Severe
* Trauma
* Ankylosing spondylitis
* Cervical pathology-related dizziness
* Spinal cord injury
* Carotid stenosis
* Other Vestibular pathologies (Meniere's disease, Vestibular hypofunction, Labyrinthitis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Dizziness | 6 weeks
  Dizziness Handicap Inventory scale (DHI) is used to assess Dizziness and can be used therapeutically to monitor and adjust rehabilitation therapy.The DHI is a 25-item self-reported measure with three categories: functional, emotional, and physical.
Quality of Life | 6 weeks
  Change in the health related quality of life using Vestibular activities and participation measure (VAP) assesses the effect of dizziness on quality of life and activities of daily living.VAP is a 34-item self-report questionnaire that asks the individual to evaluate the effect of dizziness and/or balance problems on their ability to perform activity and participation tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No